CLINICAL TRIAL: NCT06389799
Title: A Phase 2, Open Label Study of PEmigatinib and REtifanlimab in Advanced Dedifferentiated LIposarcoma
Brief Title: A Phase 2, Open Label Study of PEmigatinib and REtifanlimab in Advanced Dedifferentiated LIposarcoma (PERELI)
Acronym: PERELI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERELI; 2022-501993-21-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Dedifferentiated Liposarcoma
MeSH Terms: conditions — Liposarcoma | interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pemigatinib + Retifanlimab (Experimental): Patients will be treated with pemigatinib monotherapy for an induction phase of 6 weeks. This period is a safety measure to assess and manage adverse events of pemigatinib before start of combination treatment. Pemigatinib will be given daily as a 3-weekly cycle (2 weeks on followed by one week off) for 2 cycles. After 6 weeks, patients will receive combination treatment with retifanlimab (Q3W) and pemigatinib also as a 3-weekly cycle (2 weeks on followed by one week off).
  Interventions: Drug: Pemigatinib; Drug: Retifanlimab

INTERVENTIONS:
Drug: Pemigatinib — selective fibroblast growth factor receptor (FGFR) inhibitor, oral tablet
Drug: Retifanlimab — PD-1 inhibitor, Intravenous infusion

SUMMARY:
Dedifferentiated liposarcomas (DDLPS) are aggressive soft tissue sarcomas with no effective medical treatment options.

Immunotherapy with checkpoint inhibitors, so-called PD-1 inhibitors, have shown some effect in DDLPS in previous studies. Effect of immunotherapy can be improved by combining it with other types of tumor drugs. Medicines that inhibit signaling via the FGF receptor, so-called FGFR inhibitors, have shown a tumor-slowing effect in DDLPS in early studies. FGFR inhibitors can also induce changes that make the tumor more available to treatment with immunotherapy.

The study aims to investigate whether the combination of an FGFR inhibitor, pemigatinib, with a PD-1 inhibitor, retifanlimab can provide a tumor-slowing effect in patients with advanced DDLPS who have progressed on first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible for the study if all of the following criteria are met:

1. Be 18 years of age or above, on day of signing informed consent.
2. Must be willing and able to provide written informed consent. Written informed consent must be signed and dated before the start of specific protocol procedures.
3. Must be willing and able to conform to and comply with all protocol requirements, including, all scheduled visits, protocol procedures, and the ability to swallow oral tablets.
4. Histologically confirmed DDLPS*. Written pathology report indicating the diagnosis of DDLPS with positive MDM2 immunohistochemistry or MDM2 amplification as demonstrated by fluorescence in situ hybridization, polymerase chain reaction (PCR) or sequencing-based methods must be available.
5. Have the presence of at least 1 measurable lesion by CT per RECIST v1.1 that is considered non amenable to surgery or other curative treatments or procedures. Tumor lesions located in a previously irradiated area or in an area subjected to other loco-regional therapy are considered measurable if progression has been demonstrated in the lesion.
6. Disease relapse or radiological progression, as determined by the Investigator, within the last 6 months after at least one line of systemic treatment.

   a. Patients considered to be medically unfit for chemotherapy, as assessed by the sarcoma centre in charge of the patient's treatment, can be considered for the trial after discussion with the trial steering committee.
7. Be willing to provide tissue by core or excisional biopsy of a tumor lesion at the time points specified in the Trial Flow Chart. Archival tumor tissue can be used instead of pre-treatment biopsy. Biopsy will only be performed if the risk of complication is considered acceptable for the patient.
8. Have a performance status of 0-2 on the ECOG Performance Scale.
9. Patient must have adequate organ function as indicated by laboratory values obtained within 14 days of receiving the first dose of study drug (see study protocol)
10. Female patients of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female patients of childbearing potential must be willing to use a highly effective method of contraception, for the course of the study through 180 days after the last dose of study medication. Please refer to Section 5.3 for list of highly effective contraception.
12. Male patients must agree to use an highly effective method of contraception starting with the first dose of study therapy through 180 days after the last dose of study therapy.

Exclusion Criteria:

1. Patient has received anticancer therapy within 28 days of the first administration of study treatment, with the exception of localized radiotherapy given to a lesion not considered for RECIST measurements.
2. Toxicity of prior therapy that has not recovered to ≤ Grade 1 with the exception of

   1. Alopecia
   2. Peripheral neuropathy
   3. Anemia not requiring transfusional support
   4. Other toxicities may be considered acceptable (not an exclusion criteria) upon discussion with the Sponsor.
3. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
4. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
5. Hypersensitivity to pemigatinib or retifanlimab or any of its excipients. 6. Patients with a prior or concurrent malignant disease whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of this clinical trial are not eligible. Exceptions include, but are not limited to, patients with a history of breast cancer, requiring continued hormonal treatment (e.g. anti-estrogen or an aromatase inhibitor), patients with a history of prostate cancer, requiring continued support with luteinizing hormone- releasing hormone (LHRH) agonists, with or without androgens, basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.

7. Has known active central nervous system (CNS) metastases and/or sarcomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include sarcomatous meningitis which is excluded regardless of clinical stability.

8. Has an active autoimmune disease requiring systemic immunosuppression with corticosteroids (> 10 mg/day of prednisone or equivalent) or immunosuppressive drugs within 14 days before the first dose of study treatment.

9. Receiving chronic systemic corticosteroids (> 10 mg/day of prednisone or equivalent):

Notes:

1. Physiologic corticosteroid replacement therapy at doses > 10 mg daily of prednisone or equivalent for adrenal or pituitary insufficiency and in the absence of active autoimmune disease is permitted.
2. Participants with a condition that requires intermittent use bronchodilators, inhaled steroids, or local steroid injections may be admitted (eg, asthma or chronic obstructive pulmonary disease exacerbation).
3. Participants using topical, ocular, intra-articular, or intranasal steroids (with minimal systemic absorption) may be admitted.
4. Brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or study treatment-related standard premedication is permitted.

   10. Has a history of organ transplant, including allogeneic stem cell transplantation.

   11. Has an active infection requiring systemic antibiotics or antifungal or antiviral treatment within 7 days before first dose of study treatment.

   12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.

   13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

   14. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 180 days after the last dose of trial treatment.

   15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.

   16. Has received prior therapy with a selective FGFR inhibitor. 17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).

   18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

   19. Has received a live vaccine within 30 days of planned start of study therapy.

a. Note: COVID-19 vaccines are allowed. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

20. Has a history of calcium or phosphate homeostasis disorder or systemic mineral imbalance with ectopic calcification of soft tissues (exception: commonly observed calcifications in soft tissues such as the skin, kidney tendon, or vessel due to injury, disease, or aging in the absence of systemic mineral imbalance).

21. Use of any potent CYP3A4 inhibitors or inducers or moderate CYP3A4 inducers within 14 days or 5 half-lives (whichever is shorter) before the first dose of study drug.

22. Has current evidence of clinically significant corneal (including, but not limited to, bullous/band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjunctivitis) or retinal disorder (including, but not limited to, macular/retinal degeneration, diabetic retinopathy, retinal detachment) as confirmed by ophthalmologic examination 23. Has a history of hypovitaminosis D currently requiring supraphysiologic doses (eg, 50,000 UI/weekly) to replenish the deficiency. Vitamin D supplements are allowed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate clinical benefit of retifanlimab and pemigatinib in patients with advanced DDLPS | 2024-2028
  evaluate clinical benefit of retifanlimab and pemigatinib in patients with advanced DDLPS

SECONDARY OUTCOMES:
To further evaluate clinical efficacy of retifanlimab and pemigatinib in DDLPS | 2024-2028
To evaluate the safety and tolerability of pemigatinib and retifanlimab | 2024-2028
To evaluate impact of treatment and disease status on quality of life | 2024-2028
To evaluate the relationship between baseline and on-treatment biomarkers and clinical activity | 2024-2028

CONTACTS AND LOCATIONS:
Locations (4):
- Oslo University Hospital HF, Oslo, Norway
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Lund
  - Karolinska Universitetssjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No